CLINICAL TRIAL: NCT00632866
Title: Randomized, Double-blind, Placebo-controlled Trial of Hydroxychloroquine in Primary Sjögren's Syndrome
Brief Title: Hydroxychloroquine Versus Placebo in Primary Sjögren's Syndrome
Acronym: JOQUER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P070125-AOM 07065
Record Dates: First submitted 2008-02-29; First posted 2008-03-11 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-07

CONDITIONS: Primary Sjögren's Syndrome
Keywords: auto-immune diseases; hydroxychloroquine; primary Sjögren's syndrome; inflammatory arthritides; inflammatory rheumatic diseases; dryness; joint diseases
MeSH Terms: conditions — Joint Diseases | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Active treatment : Hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine : 200mg / day since 24 weeks
  Other Names: Plaquenil
  Arms: 1
Drug: Placebo — Placebo : 2cp/ day since 24 weeks
  Arms: 2

SUMMARY:
Primary Sjögren's syndrome (SJp) affects 0.1% of the population. This systemic autoimmune disease systemic is characterized by disabling dryness, fatigue and pain, and systemic complications in 30% of patients. No treatment has proven effective in this disease. In open studies, some efficacy was observed with hydroxychloroquine but no RCT versus placebo has ever been done.

Thus, the primary purpose of this study is to evaluate the efficacy and safety of hydroxychloroquine (400mg/ day) on dryness, pain, and fatigue, assessed by the patient using visual analogical scales.

DETAILED DESCRIPTION:
Primary Sjögren's syndrome (SJp) affects 0.1% of the population. This systemic autoimmune disease systemic is characterized by disabling dryness, fatigue and pain, and systemic complications in 30% of patients. No treatment has proven effective in this disease. In open studies, some efficacy was observed with hydroxychloroquine but no RCT versus placebo has ever been done.

Thus, the primary purpose of this study is to evaluate the efficacy and safety of hydroxychloroquine (400mg/ day) on dryness, pain, and fatigue, assessed by the patient using visual analogical scales (VAS).

Response is defined by the improvement of 30% or more of at least 2 out of 3 of the following VAS : most disabling dryness, fatigue, and pain.

ELIGIBILITY:
Inclusion criteria:

* Patients suffering from primary Sjögren's syndrome according to the European-American consensus group criteria
* Male and female aged of 18 or more
* Conducting a clinical examination beforehand.
* Having undergone less than 6 months before an ophthalmological examination, which did not counter-indicated hydroxychloroquine.
* Patient without heart conduction disturbance (PR>=0.2 sec and QRS>=0.08 sec).
* Patient with the ability to give informed, dated and signed consent before the beginning of any proceedings related to the trial
* Patients treated with corticosteroids and / or NSAIDs, and / or cyclosporine, and / or pilocarpine must have received stable doses of these treatments during the month preceding inclusion.

Exclusion criteria:

* SJ associated with other autoimmune diseases
* Retinopathy /severe cataract/ monophthalmos
* Previous or ongoing treatment by hydroxychloroquine
* Treatment by another immunosuppressant not interrupted at least 4 weeks prior to inclusion, or 6 months prior to inclusion for cyclophosphamide or rituximab
* lymphoma or other severe SJp complications: vasculitis responsible for a documented renal, neurological, digestive or heart involvement, glomerular disease associated with hematuria and / or proteinuria > 0.5 g / d), CNS involvement, peripheral neurological involvement with motor deficiency scored at 3 or less on a scale of 5 , interstitial pneumonitis, recent symptomatic cryoglobulinemia with neurological, renal, or other systemic involvement, myositis with motor deficiency (isolated purpura is not an exclusion criteria)
* Chronic Alcoholism
* Hepato-cellular insufficiency
* Creatinine clearance <60 ml / min
* Risk of lost follow-up
* People younger than 18, major trusteeship and guardianship, or deprived of liberty
* Pregnancy /Breastfeeding
* Hypersensitivity to chloroquine or to hydroxychloroquine or any of the other constituents of Plaquenil
* Psoriasis or intermittent porphyria.
* G6PD deficiency, congenital galactosemia, malabsorption syndrome, glucose and galactose, or lactase deficiency.
* Non-membership in a social security system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2008-03; Primary Completion 2011-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an improvement of 30% or more of at least 2 out of the 3 following VAS: 1. the most disabling dryness 2. pain 3. fatigue | 6 months

SECONDARY OUTCOMES:
SCHIRMER's test, van BIJSTERVELD score, salivary flow, disease systemic features, quality of life, interferon-inducible genes expression Association between clinical response and hydroxychloroquine blood level, interferon-inducible genes expression | 6 mois

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Bicëtre, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Gottenberg JE, Ravaud P, Puechal X, Le Guern V, Sibilia J, Goeb V, Larroche C, Dubost JJ, Rist S, Saraux A, Devauchelle-Pensec V, Morel J, Hayem G, Hatron P, Perdriger A, Sene D, Zarnitsky C, Batouche D, Furlan V, Benessiano J, Perrodeau E, Seror R, Mariette X. Effects of hydroxychloroquine on symptomatic improvement in primary Sjogren syndrome: the JOQUER randomized clinical trial. JAMA. 2014 Jul 16;312(3):249-58. doi: 10.1001/jama.2014.7682. PMID 25027140